CLINICAL TRIAL: NCT03283436
Title: Superior Hypogastric Plexus Block During Laparoscopic Hysterectomy: a Randomized Controlled Trial.
Brief Title: RCT Superior Hypogastric Block During LH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jon I. Einarsson (Other)
Collaborators: University of North Carolina (Other); George Washington University (Other)
Responsible Party: Sponsor-Investigator, Jon I. Einarsson, Division Chair, Minimally Invasive Gynecology, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017P001804
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Hysterectomy
Keywords: Laparoscopy; Superior hypogastric plexus block
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded to the treatment arm; however, the surgeon will know if a patient has been randomized to receive the block during the hysterectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Superior hypogastric plexus block (Experimental): Prior to the laparoscopic hysterectomy and any additional procedures, the SHPB will be performed on patients in the treatment arm. The block will contain 10 mL of 0.25% bupivacaine hydrochloride (Bupivacaine; 2.5 mg/mL = 25 mg). The anesthetic works by blocking nerve conduction and the steroid by reducing inflammation. The injection will be performed by tenting the presacral peritoneum, aspirating with a laparoscopic needle-tip syringe to ensure extravascular placement, and injecting the block.
  Interventions: Drug: Bupivacaine Hydrochloride 0.25% Injection Solution
- No block (No Intervention): Patients in the control arm will undergo the hysterectomy with no intervention.

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride 0.25% Injection Solution — 10 mL of 0.25% bupivacaine hydrochloride (2.5 mg/mL = 25 mg)
  Other Names: Bupivacaine
  Arms: Superior hypogastric plexus block

SUMMARY:
The goal of this study is to assess the efficacy of a superior hypogastric plexus block (SHPB) for pain relief following a laparoscopic hysterectomy.

DETAILED DESCRIPTION:
The objective of this study is to assess the efficacy of a SHPB for pain relief following laparoscopic hysterectomy. The superior hypogastric plexus lies in the presacral space and supplies autonomic innervation to the central pelvis. This plexus is suspected to play a role in postoperative pain following a hysterectomy. The investigators hypothesize that a SHPB using the anesthetic bupivacaine will reduce patients' pain scores and opioid consumption following a laparoscopic hysterectomy. Intraoperative and immediate postoperative opioid consumption will be collected from the Medication Administration Record by the nursing staff. The nursing staff will also be asked to complete a recovery worksheet that details the Visual Analog Scale pain score and opioid administration on admission to the recovery unit and every postoperative hour until six hours or the patient is discharged. Patients will also be asked to complete a daily diary for one week following the procedure, which details their pain level and daily opioid consumption. Patients will be followed for thirty days after surgery to assess for the occurrence of any postoperative complications. Detailed patient and procedure characteristics including age, race, body mass index, parity, surgical history, surgery indication, procedure type, and surgical approach will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18
* English Speaking
* Able to provide informed consent
* Undergoing laparoscopic hysterectomy for benign indications

Exclusion Criteria:

* Planned laparotomy incision
* Planned procedure that requires dissection of the presacral space
* Allergy to block medication (s)
* Known or suspected malignancy
* Non-English speaker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Clark NV, Moore K, Maghsoudlou P, North A, Ajao MO, Einarsson JI, Louie M, Schiff L, Moawad G, Cohen SL, Carey ET. Superior Hypogastric Plexus Block to Reduce Pain After Laparoscopic Hysterectomy: A Randomized Controlled Trial. Obstet Gynecol. 2021 Apr 1;137(4):648-656. doi: 10.1097/AOG.0000000000004329. PMID 33706344

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Superior Hypogastric Plexus Block | No Block
Started | 50 | 50
Completed | 44 | 50
Not Completed | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Superior Hypogastric Plexus Block | No Block | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [40 to 48] | 45 [41 to 49] | 45 [41 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White/Caucasian | 35 | 29 | 64
  Race/Ethnicity: Black/African American | 8 | 14 | 22
  Race/Ethnicity: Hispanic | 2 | 2 | 4
  Race/Ethnicity: Asian | 2 | 2 | 4
  Race/Ethnicity: Other | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 28.7 [24.2 to 33.2] | 30.5 [25.4 to 35.6] | 29.5 [24.4 to 34]
Gravidity [Median (Inter-Quartile Range); unit: Pregnancies] | 2 [0.5 to 3.5] | 2 [0.5 to 3.5] | 2 [0.5 to 3.5]
Parity [Median (Inter-Quartile Range); unit: Pregnancies] | 2 [1.5 to 2.5] | 2 [0.5 to 3.5] | 2 [1 to 3]
Indication for Surgery [Count of Participants; unit: Participants]
  Fibroids | 25 | 20 | 45
  Abnormal Uterine Bleeding | 10 | 13 | 23
  Pelvic pain | 12 | 16 | 28
  Other | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Scores
Description: The primary outcome will be immediate postoperative patient pain scores using the Visual Analog Scale (VAS) in the recovery unit. Postoperative pain scores will be collected every one hour, on a scale from 1 to 10. Higher score indicates greater pain intensity. The score reported here is the mean VAS score in the first 2 hours.
Time Frame: Admission to recovery unit and every hour after for 2 hours
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Superior Hypogastric Plexus Block | No Block
Number analyzed (Participants) | 50 | 50
score on a scale | 3.9 [1.6 to 6.3] | 4.7 [3.2 to 6.2]

2. Secondary Outcome: Postoperative Opioid Use
Description: Patients will be asked to complete a daily diary for one week that records their daily postoperative opioid consumption.
Time Frame: Admission to recovery unit to 1 week post op, assessed up to 1 week after surgery
Measure: Median (Inter-Quartile Range); unit: milligrams morphine equivalents
Arm/Group | Superior Hypogastric Plexus Block | No Block
Number analyzed (Participants) | 50 | 50
milligrams morphine equivalents
  postoperative day 0 | 5 [-1.9 to 11.9] | 10.2 [4 to 16.5]
  postoperative day 1 | 2.5 [0 to 5] | 5 [0 to 10]
  postoperative day 2 | 0 [-2.5 to 2.5] | 2.5 [0 to 5]
  postoperative day 3 | 0 [-1.3 to 1.3] | 3.5 [1 to 6]
  postoperative day 4 | 0 [-1.3 to 1.3] | 0 [-1.3 to 1.3]
  postoperative day 5 | 0 [0 to 0] | 0 [0 to 0]
  postoperative day 6 | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Postoperative Pain Scores
Description: Patients will be asked to complete a daily diary for one week following the procedure, which details their pain level using VAS pain scores from the Brief Pain Inventory (BPI). Pain is reported on a scale of 1 to 10, and a higher score indicates greater pain intensity.
Time Frame: Discharge to 1 week after surgery, assessed up to 1 week after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Superior Hypogastric Plexus Block | No Block
Number analyzed (Participants) | 50 | 50
score on a scale
  postoperative day 0 | 5 [2.3 to 7.8] | 6 [4.6 to 7.4]
  postoperative day 1 | 6.3 [4.5 to 8.1] | 5.6 [4.2 to 7]
  postoperative day 2 | 5.5 [3.6 to 7.5] | 5 [3.9 to 6.2]
  postoperative day 3 | 4.1 [2.4 to 5.8] | 4 [2.6 to 5.4]
  postoperative day 4 | 4 [2.3 to 5.7] | 4 [2.5 to 5.5]
  postoperative day 5 | 3 [1.5 to 4.6] | 3.5 [2.3 to 4.8]
  postoperative day 6 | 2.8 [1.3 to 4.4] | 2.8 [1.6 to 4.1]

ADVERSE EVENTS:
Time Frame: one month after surgery for each study participant
Arm/Group | Superior Hypogastric Plexus Block | No Block
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT03283436/Prot_SAP_000.pdf